CLINICAL TRIAL: NCT06864728
Title: The Impact of Social Determinates of Health on Risk for Diabetes in the Hispanic Community: a Pilot Study
Brief Title: Diabetes Prevention in Hispanic Adults Using Constant Glucose Monitors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00005535
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Prediabetes / Type 2 Diabetes
Keywords: diabetes risk; constant glucose monitoring; diabetes knowledge
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: No additional details.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In Person patient education (Active Comparator): Participants will receive patient education in person or virtually. They will get the results from their tests
  Interventions: Behavioral: In person or virtual diabetes education
- Video Intervention (Experimental): Patients will receive a link to a video of a nurse explaining their results.
  Interventions: Behavioral: Video Diabetes Education

INTERVENTIONS:
Behavioral: Video Diabetes Education — Participants will receive a link to a short video explaining their findings. They can use the link as often as they'd like. They will get the results for the CGM and the laboratory findings. They will be linked to their 2 week diet diary
  Arms: Video Intervention
Behavioral: In person or virtual diabetes education — Participants will meet with a nurse to discuss their CGM results and their lab results and get appropriate education.
  Arms: In Person patient education

SUMMARY:
The purpose of the study is twofold: to see the impact of your environmental stress on daily glucose changes and to create an intervention using CGM to potentially decrease risk for diabetes. The aim of this study to develop an intervention to prevent diabetes in the Hispanic community and inform policies about social determinants of health.

DETAILED DESCRIPTION:
Social determinants of health are associated with developing diabetes mellitus type 2 (diabetes) onset, progression, and adverse outcomes. Hispanics have a 50% lifetime risk of developing diabetes. They also transition from pre-diabetes to diabetes faster and have an earlier onset of diabetes and its complications than the general population. People with a family history of diabetes are 7.6 times more likely to develop diabetes than individuals without such a history. Diabetes research uses hemoglobin A1C (A1C), the accumulation of glucose on hemoglobin molecules during the past three months, as the measure of diabetes control. However, A1C is an insensitive measure of glucose for those at risk for developing diabetes because glucose spikes and variability are often masked in an average glucose level by A1C. Glucose spikes should rarely occur and can be an early indicator of insulin insufficiency. Constant glucose monitors (CGM) can detect glucose spikes and have successfully lowered A1C in people with diabetes.

Using CGM, Hispanic adults with familial risk factors of diabetes can obtain a more detailed assessment of their glucose levels and identify foods, activities, emotions, and stress that impact their glucose levels. Time constraints can often be a barrier to participating in an intervention. The proposed intervention will test an asynchronous nurse-led intervention. To address this gap and create an intervention, glucose variability in Hispanics at risk for diabetes will be investigate to identify glucose variability predictors and create a culturally tailored intervention to prevent diabetes.

Diagnosis of glucose intolerance, or prediabetes, can be evaluated using an oral glucose tolerance test (oGTT) to illustrate a person's ability to produce and use insulin in response to glucose consumption. The medical community uses these lab values as benchmarks. Knowing the starting level of participants' glucose tolerance will allow us to better interpret the CGM findings. Additionally, it will provide validity for using CGMs in the population at risk for diabetes.

Therefore, the specific aims are as follows:

1. To examine the relationship between social determinants and glucose control. These analyses estimate the associations between economic instability, neighborhood vulnerability, food insecurity, and healthcare quality with glucose variability.
2. To determine the feasibility and acceptability of a CGM intervention for Hispanics at risk of diabetes. The study compares synchronous or asynchronous diabetes education intervention. The participants will receive education and feedback based on their CGM results, either in person or via videos.

ELIGIBILITY:
Inclusion Criteria:

* self- identify as Hispanic Has a parent diagnosed with diabetes type 2

Exclusion Criteria:

* Pregnant Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Diabetes Knowledge | 4 weeks
  measured by the Diabetes Knowledge questionnaire - Revised

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be deidentified. Formal request to the PI of the study will be considered.